CLINICAL TRIAL: NCT00691821
Title: A 12-week, Prospective, Open-label, Randomized, Controlled Clinical Trial Comparing Negative Pressure Wound Therapy (NPWT) to Standard Wound Care for the Treatment of Chronic Pressure Wounds of the Pelvic Region
Brief Title: Negative Pressure Wound Therapy for the Treatment of Chronic Pressure Wounds
Acronym: NPWT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Patients not meeting inclusion criteria, therefore recruitment rate low, terminated due to the lack of feasibility to complete the study in a timely manner.
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government); Unity Health Toronto (Other); Women's College Hospital (Other); Hamilton Niagara Haldimand Brant Community Care Access Centre (Other); Toronto Central Community Care Access Centre (Other)
Responsible Party: Ron Goeree, MA Director of PATH Research Institute, St. Joseph's Healthcare Hamilton, Associate Professor, Department CE&B, McMaster University, Programs for Assessment of Technology in Health (PATH) Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HTA012-0801-01
Record Dates: First submitted 2008-05-27; First posted 2008-06-05 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2011-07

CONDITIONS: Skin Ulcer; Pressure Ulcer
Keywords: Negative-Pressure Wound Therapy; Bandages; Community Health Services
MeSH Terms: conditions — Skin Ulcer; Pressure Ulcer | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Standard Dressings
  Interventions: Other: Standard Dressings
- 2 (Experimental): Negative Pressure Wound Therapy
  Interventions: Device: Negative Pressure Wound Therapy (Vacuum-Assisted Closure System [V.A.C.® Therapy™, KCI Medical Canada Inc., Mississauga, Ontario])

INTERVENTIONS:
Other: Standard Dressings — Participants will receive standard dressings changes as needed. Different dressing types (e.g., silver, simple gauze, hydrogel, foam, creams, gels) will be used dependent on the type of the wound (e.g., dry, wet, and intermediate).
  Arms: 1
Device: Negative Pressure Wound Therapy (Vacuum-Assisted Closure System [V.A.C.® Therapy™, KCI Medical Canada Inc., Mississauga, Ontario]) — Participants will receive negative pressure wound therapy.
  Other Names: V.A.C. Therapy
  Arms: 2

SUMMARY:
The purpose of this study is to assess the difference in the percent reduction in wound surface area, without surgery, of chronic pressure ulcers of the pelvic region for Negative Pressure Wound Therapy (NPWT) compared to the standard dressing. This study is designed to provide evidence regarding NPWT as compared to standard dressing regimens and compare the efficacy, safety, effectiveness and cost-effectiveness.

DETAILED DESCRIPTION:
The Ontario Health Technology Advisory Committee recommended that a study should be completed due to the large numbers of patients needing chronic wound care and the increasing use of NPWT based on poor quality evidence to identify any potential indications for the use of NPWT. This study is designed to provide evidence regarding NPWT as compared to standard dressing regimens in Ontario and the results will serve as a benchmark for the utilization of NPWT in chronic pressure wounds, establishing and providing guidance regarding the use of NPWT in this population of subjects and to support policy decision making regarding the funding of the NPWT in the province. Specifically, this will compare the efficacy, effectiveness and cost-effectiveness of NPWT with standard dressing regimens for the treatment of chronic pressure ulcers of the pelvic region.

This is a prospective, randomized, open-label, controlled clinical trial comparing standardized wound dressing (control arm) to NPWT (experimental arm) for the treatment of chronic pressure wounds of the pelvic region. NPWT will be performed using the Vacuum-Assisted Closure System (V.A.C.® Therapy™, KCI Medical Canada Inc., Mississauga, Ontario). NPWT will be compared to the present recommended state of the art wound dressings in subjects who would be candidates for either type of wound therapy. Both arms will receive standard wound care (e.g., debridement, preventative care, infection control, etc.). The efficacy, effectiveness, safety, and quality of life will be evaluated for standardized wound dressing versus NPWT. Complications associated with either form of wound care will be documented. An economic evaluation will be conducted in order to assess the cost-effectiveness and cost-utility of NPWT compared to standard wound dressing. It is anticipated that 184 subjects will be enrolled and randomized over a 1.5 year period. All subjects providing consent and meeting inclusion/exclusion criteria will be randomized to either treatment arm and followed for 12 weeks. Patients who have wound closure within the 12-week study period will continue to have wound care visits as scheduled. All subjects will have Wound Evaluation Visits and Wound Dressing Change Visits. Wound Evaluation Visits will occur at baseline, 2, 4, 6, 8 and 12 weeks after the date of randomization, where following removal of the dressing, a detailed wound assessment (e.g., wound characteristics, measurements) will be done and healthcare resource utilization will be collected. Disease specific quality of life measures and preference based quality of life measures (EQ-5D) will be collected at baseline, 6 weeks and at 12 weeks. Dressing Change Visits will occur as clinically required and the frequency of dressing changes per week will be allowed to vary over the 12 weeks of the study. During the dressing change visits, subjects will be monitored for wound infection and other complications. Subjects may be enrolled and randomized in the clinic and transferred to the community with continued follow-up completed by the appropriate Community Care Access Centre.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. All chronic pressure wounds of the pelvic region except trochanteric wounds.
3. Chronic pressure wound defined as the presence of a pressure wound for > 6 weeks and < 6 months with no sign of improvement in healing
4. Wound size surface area > 2cm2
5. Stage III-IV pressure ulcer according to the National Pressure Ulcer Advisory Panel (NPUAP)
6. No clinical signs of active infection at the wound site and currently not on antibiotics
7. Willingness to off-load or pressure redistribute ulcer

Exclusion Criteria:

1. Candidate for surgery in the next 12 weeks
2. A wound with necrotic tissue unable to tolerate debridement
3. Exposed blood vessels and/or organs within the wound
4. Chronic osteomyelitis (as determined by biopsy) or osteomyelitis that is not treatable by debridement and antibiotics
5. Non-enteric or unexplored fistulae
6. Wounds requiring hemostasis (i.e., that the flow of blood be stopped) for local bleeding
7. Alternate etiology for non-healing
8. Concomitant conditions that in the judgment of the investigator would make the subject inappropriate for entry to the study (e.g., malignancy in wound, malignancy less than 1-year disease free interval, previous or current irradiation, known immunodeficiency and/or major uncorrected medical disorders such as serious non-malignant disease, serious cardiovascular or pulmonary disease, lupus, inflammatory bowel disease, palliative care or sickle cell disease)
9. Poor nutritional status as determined by a Braden Scale Nutritional Assessment score of 2 or 1 with a serum albumin < 25 g/L and hemoglobin < 90 g/L
10. Currently taking medication that may interfere with wound healing (e.g., oral systemic steroids, immunosuppressive drugs, unfractionated heparin infusion)
11. Women who are currently pregnant or are breast feeding; or women of child bearing potential who are not currently taking adequate birth control
12. Participation in another investigative drug or device trial currently or within the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the percent reduction in wound surface area, without surgery, at 12 weeks compared to wound measurements at treatment initiation following randomization. | 12 Weeks

SECONDARY OUTCOMES:
Wound healing, effectiveness, safety, healthcare resource utilization, costing, quality of life, cost effectiveness analysis | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ron Goeree, MA, Study Chair — Programs for Assessment of Technology in Health Research Institute; James Mahoney, MD, Principal Investigator — Unity Health Toronto; Gary Sibbald, MD, Principal Investigator — Women's College; Maureen Kitson, Principal Investigator — Niagara Region Community Care Access Centre; Joanne Greco, BScN, Principal Investigator — Toronto Central Community Care Access Centre
Locations (4):
- Canada (4):
  - Niagara Branch - Hamilton Niagara Haldimand Brant Community Care Access Centre, Saint Catherines, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Women's College Hospital, Toronto, Ontario
  - Toronto Central Community Care Access Centre, Toronto, Ontario